CLINICAL TRIAL: NCT06742099
Title: Outcome of Intercostal Tube Insertion and Pleurodesis for Malignant Pleural Effusion
Brief Title: The Outcome of Inserting Intercostal Tube or Pleurodesis for Malignant Pleural Effusion
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hussein Essameldin Hussein Mohamed, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICT Malignant Pleural effusion
Record Dates: First submitted 2024-12-05; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Malignant Pleural Effusions (Mpe)
MeSH Terms: conditions — Pleural Effusion, Malignant; Myeloproliferative Disorder, Chronic, with Eosinophilia | interventions — Pleurodesis

STUDY DESIGN:
Intervention Model Description: 2.4.1- Type of the study: Retrospective and Prospective 2.4. 2- Study Setting: All patients with malignant pleural effusion and either underwent intercostal tube insertion or had pleurodesis done in 2 to 3 years' timeframe.
  2.4. 3- Study subjects:
  1. Inclusion criteria:
     All patients presented with malignant pleural effusion to Assiut University Hospital regardless of sex And age
  2. Exclusion criteria:
     All patients presented with pleural effusion other than malignant pleural effusion, including patients with debilitating diseases and terminal patients.
  3. Sample Size Calculation:
  Sample size calculation was carried out using G* Power 3 software. To detect significant differences between both groups as regard post-operative complications with expected frequency of 14.5-16.7% and based on the following parameters: an error probability of 0.05 and 80% power on a two-tailed test, a calculated minimum required sample of 110 patients will be required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Malignant Pleural effusion with pleurodesis (Active Comparator): these are patients who have malignant pleural effusion and will have talc injected into the pleural cavity to induce pleurodesis
  Interventions: Procedure: Intercostal chest tube; Combination Product: Pleurodesis
- Malignant Pleural effusion with only chest tube for drainage (Active Comparator): these are patients who have malignant pleural effusion but will only have intercostal chest tube inserted for drainage
  Interventions: Procedure: Intercostal chest tube

INTERVENTIONS:
Procedure: Intercostal chest tube — the use of chest tubes to drain malignant pleural effusion
  Other Names: Pleurodesis
Combination Product: Pleurodesis — the injection of Talc in pleural space to induce inflammation reaction and produce pleurodesis
  Arms: Malignant Pleural effusion with pleurodesis

SUMMARY:
Approximately half of all patients with metastatic cancer develop a malignant pleural effusion which is likely to lead to a significant reduction in quality of life secondary to symptoms such as dyspnoea and cough. The aim of pleurodesis in these patients is to prevent re-accumulation of the effusion and thereby of symptoms,and avoid the need for repeated hospitalization for thoracocentesis. Numerous clinical studies have been performed to try to determine the optimal pleurodesis strategy, and synthesis of the available evidence should facilitate this. The treatment of MPE is aimed at palliating symptoms since no intervention has been shown to improve survival in this population and since survival is generally limited in cancers that have spread to the pleural space. In this palliative setting, only patients symptomatic from their MPE should be submitted to further intervention. As well, further interventions in symptomatic patients should be limited to those patients who have experienced symptomatic improvement following initial therapeutic thoracentesis. The two main treatment approaches to MPE are to obliterate the pleural space via a pleurodesis procedure or to chronically drain the pleural cavity with Intercostal tube. The aims of this review were to ascertain the optimal procedure in cases of malignant pleural effusion in terms of patients' quality of life post procedure, recurrence of effusion.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented with malignant pleural effusion to Assiut University Hospital regardless of sex and age

Exclusion Criteria:

* All patients presented with pleural effusion other than malignant pleural effusion, including patients with debilitating diseases and terminal patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
chest imaging, chest x-rays will be used to record the progress of the malignant pleural effusion in both treatments | from the time of intervention up to 6 months
  efficacy of both treatments, in which the treatment that shows less accumulation of pleural effusion in chest imaging gets better results hence is more effective than the other in terms of reducing Malignant Pleural effusion
A questionnaire will be used to assess tolerability of both treatments on patients | from the time of intervention up to 6 months
  Tolerability, in which the questionnaire will include a score from 1 to 10 in which 1 is the lowest point and 10 is the highest point, it will include how painful each treatment is and how quality of life has changed after each treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beltsios ET, Mavrovounis G, Adamou A, Panagiotopoulos N. Talc pleurodesis in malignant pleural effusion: a systematic review and meta-analysis. Gen Thorac Cardiovasc Surg. 2021 May;69(5):832-842. doi: 10.1007/s11748-020-01549-2. Epub 2020 Nov 22. PMID 33222091
- [Background] Bhatnagar R, Piotrowska HEG, Laskawiec-Szkonter M, Kahan BC, Luengo-Fernandez R, Pepperell JCT, Evison MD, Holme J, Al-Aloul M, Psallidas I, Lim WS, Blyth KG, Roberts ME, Cox G, Downer NJ, Herre J, Sivasothy P, Menzies D, Munavvar M, Kyi MM, Ahmed L, West AG, Harrison RN, Prudon B, Hettiarachchi G, Chakrabarti B, Kavidasan A, Sutton BP, Zahan-Evans NJ, Quaddy JL, Edey AJ, Clive AO, Walker SP, Little MHR, Mei XW, Harvey JE, Hooper CE, Davies HE, Slade M, Sivier M, Miller RF, Rahman NM, Maskell NA. Effect of Thoracoscopic Talc Poudrage vs Talc Slurry via Chest Tube on Pleurodesis Failure Rate Among Patients With Malignant Pleural Effusions: A Randomized Clinical Trial. JAMA. 2020 Jan 7;323(1):60-69. doi: 10.1001/jama.2019.19997. PMID 31804680
- [Background] Toth JW, Reed MF, Ventola LK. Chest Tube Drainage Devices. Semin Respir Crit Care Med. 2019 Jun;40(3):386-393. doi: 10.1055/s-0039-1694769. Epub 2019 Sep 16. PMID 31525813